CLINICAL TRIAL: NCT01756326
Title: A Pivotal Phase 2b/3, Multicentre, Randomised, Open, Controlled Study on the Efficacy and Safety of Autologous Osteoblastic Cells (PREOB®) Implantation in Non-Infected Hypotrophic Non-Union Fractures
Brief Title: Study on Autologous Osteoblastic Cells Implantation in Hypotrophic Non-Union Fractures
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: focus resources in the allogeneic platform and provide optimal value for patients
Sponsor: Bone Therapeutics S.A (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PREOB-NU3
Record Dates: First submitted 2012-12-20; First posted 2012-12-25 (Estimated); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Long Bone Non-Union
Keywords: Non-Union Fractures; Impaired Healing; Fractures; Orthopedics; Bone; Musculoskeletal Disorders
MeSH Terms: conditions — Fractures, Bone; Musculoskeletal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PREOB® Implantation (Experimental): Each patient will undergo a single administration of PREOB® into the non-union site, under local or loco-regional anesthesia.
  Interventions: Drug: PREOB® Implantation
- Bone Autograft (Active Comparator): Each patient will be treated by Bone Autograft according to standard-of-care procedure of the investigating site.
  Interventions: Procedure: Bone Autograft

INTERVENTIONS:
Drug: PREOB® Implantation
  Arms: PREOB® Implantation
Procedure: Bone Autograft
  Arms: Bone Autograft

SUMMARY:
Fracture healing is a complex physiological process caused by interaction of cellular elements, cytokines and signaling proteins, which results in the formation of new bone (Gerstenfeld et al., 2003). Depending on fracture site, complexity, co-morbidities and other factors, 10% of all fractures will eventually fail to unite.

Non-union fractures are defined as fractures that are at least six to nine months old and in which there have been no signs of healing for the last three months. Various causes have been evoked for impaired healing in hypotrophic (atrophic and oligotrophic) non-unions, including poor fracture stabilization, local infection and failure of the osteoblastic cells to multiply. Currently the treatment of choice for non-unions, particularly atrophic non-unions, is bone autograft (or allograft), combined or not with intramedullary nailing, plating, and external fixation devices (Kanakaris et al., 2007). This procedure produces good results but requires an invasive surgery of several hours under general anesthesia and a few days of hospitalization. Because of this, major complications have been reported in up to 20-30% of patients (Pieske et al., 2009, Zimmerman et al., 2009).

This Phase 2b/3 study aims at demonstrating the safety and efficacy of PREOB®, a proprietary population of autologous osteoblastic cells, in the treatment of hypotrophic non-union fractures of long bones. PREOB® will be compared to Bone Autograft in a non-inferiority design.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide a written, dated, and signed informed consent prior to any study related procedure, and to understand and comply with study requirements
* Diagnosis of a non-infected hypotrophic non-union fracture of a long bone of at least 6 months at the time of treatment
* Normal hematology function

Exclusion Criteria:

* Positive serology for HIV, hepatitis B, hepatitis C, syphilis, HTLV-1
* Presence or previous history, or risk factors for diseases caused by prions
* Renal impairment, hepatic impairment
* Patient with poorly controlled diabetes mellitus, severe arterial diseases and/or neuropathy
* Insufficient fracture stability
* Recent osteosynthesis material or bone graft
* Multifocal fracture/non-unions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-06; Primary Completion 2018-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Global Disease Evaluation as perceived by the patient using a Visual Analogue Scale | 12 months
Radiological healing progression using the RUS(T) as assessed by CT scan | 12 months
Potential occurrence of any AE or SAE, related to the product or to the procedure, using patient open non-directive questionnaire, physical examination and laboratory measurements | 12 months

SECONDARY OUTCOMES:
Pain using a Visual Analogue Scale | 12 months
Weight-bearing using Likert Scale | 12 months
Well-being score as assessed by the SF-12 questionnaire | 12 months
Radiological improvement using the RUS(T) as assessed by X-ray | 12 months

CONTACTS AND LOCATIONS:
Locations (16):
- Belgium (9):
  - Investigating site BE01, Anderlecht
  - Investigating site BE05, Bruges
  - Investigating site BE09, Brussels
  - Investigating site BE02, Charleroi
  - Investigating site BE04, Genk
  - Investigating site BE06, Ghent
  - Investigating site BE07, Hasselt
  - Investigating site BE08, Mons
  - Investigating site BE03, Ottignies
- France (5):
  - Investigating site FR01, Amiens
  - Investigating site FR04, Bordeaux
  - Investigating site FR06, Évry
  - Investigating site FR03, Paris
  - Investigating site FR02, Rouen
- Netherlands (2):
  - Investigating site NL02, Maastricht
  - Investigating site NL01, Rotterdam